CLINICAL TRIAL: NCT01897038
Title: A Phase Ib, Open-Label Study Evaluating The Safety, Tolerability, and Pharmacokinetics of Onartuzumab Given as a Single Agent and in Combination With Sorafenib in Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: A Safety, Tolerability, and Pharmacokinetics Study of Onartuzumab as Single Agent or in Combination With Sorafenib in Participants With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO28651
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — onartuzumab; Sorafenib

ARMS (2):
- Cohort 1 (Onartuzumab) (Experimental)
  Interventions: Drug: Onartuzumab
- Cohorts 2/3 (Onartuzumab + Sorafenib) (Experimental)
  Interventions: Drug: Onartuzumab; Drug: Sorafenib

INTERVENTIONS:
Drug: Onartuzumab — Onartuzumab intravenous infusion at a starting dose of 10 or 15 milligram per kilogram body weight administered every 3 weeks (Q3W) until disease progression or unacceptable toxicity occurs (maximum up to 31 months).
  Other Names: RO5490258
Drug: Sorafenib — Sorafenib 400 milligram (mg) tablets (2 tablets of 200 mg each) orally once daily or twice daily depending on the cohort assigned until disease progression or unacceptable toxicity occurs (maximum up to 31 months).
  Arms: Cohorts 2/3 (Onartuzumab + Sorafenib)

SUMMARY:
This multicenter, open-label study will evaluate the maximum tolerated dose (MTD) and dose-limiting toxicities of onartuzumab as single agent or in combination with sorafenib in participants with advanced hepatocellular carcinoma. Participants in Cohort 1 will receive onartuzumab as single agent on Day 1 of each 21-day cycle. Participants in Cohorts 2 or 3 will receive onartuzumab on Day 1 of each 21-day cycle in combination with sorafenib 400 mg orally daily or twice daily. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Cytologically or histologically confirmed diagnosis of hepatocellular carcinoma (HCC)
* Advanced or metastatic disease
* Not a candidate for curative treatments (that is, resection, transplantation)
* Child-Pugh class A liver function
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Life expectancy greater than (>) 3 months
* For participants who received prior adjuvant chemotherapy, a treatment-free interval of at least 6 months between the last chemotherapy cycle and Cycle 1 Day 1

Exclusion Criteria:

* Prior surgery or local therapy within 4 weeks prior to Cycle 1 Day 1, with the exception of palliative radiation therapy to the bone
* Brain metastasis or spinal cord compression not definitively treated with surgery and/or radiation
* Granulocyte count less than (<) 1500 per cubic millimeter (mm^3), platelet count < 75,000/mm^3, and hemoglobin < 8 gram per deciliter (g/dL) within 7 days prior to Cycle 1 Day 1
* Total bilirubin greater than (>) 1.5 times the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT), Alanine transaminase (ALT) serum glutamic-pyruvic transaminase (SGPT), alkaline phosphatase (ALP) > 5 × ULN
* Serum creatinine > 1.5 × ULN or creatinine clearance < 60 cubic centimeter per minute (cc/min) by Cockcroft-Gault formula
* Significant history of cardiac disease within 6 months prior to Cycle 1 Day 1, myocardial infarction within the previous year, or current cardiac ventricular arrhythmias requiring medication
* Serious active infection, or other serious underlying medical conditions that would impair the ability of the participant to receive protocol treatment, with the exception of hepatitis B virus (HBV) and hepatitis C virus (HCV) infections
* Known active infection with human immunodeficiency virus (HIV) or known HIV-seropositivity
* Inability to take oral medication or untreated malabsorption syndrome
* Pregnant or lactating women
* History of transplantation including organ, bone marrow transplantation, and peripheral blood stem cell transplantation with the exception of corneal transplantation
* Active bleeding diathesis (including active esophageal varices) or tumor rupture within 8 weeks prior to Cycle 1 Day1 that are not successfully treated
* Uncontrolled hypertension
* Treatment with any other investigational drug within 4 weeks of Cycle 1 Day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLT) | Maximum up to 42 days
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | Up to approximately 31 months

SECONDARY OUTCOMES:
Area Under the Concentration-time Curve (AUC) of Onartuzumab | Day 1 up to Day 15 of Cycle 1, Day 1 of Cycle 2, 3, 4, and every fourth cycle thereafter (maximum up to 31 months)
Steady-state Plasma Concentrations of Sorafenib When Administered in Combination With Onartuzumab | Day 1 Cycles 1-2
Progression-free Survival (PFS) | Up to approximately 31 months
Percentage of Participants With Objective Response | Up to approximately 31 months
Duration of Response (DR) | Up to approximately 31 months
Overall Survival (OS) | Up to approximately 31 months
Percentage of Participants With Progression-free Survival at 4 Months (PFS4) | 4 months
Number of Participants With Anti-therapeutic Antibodies (ATAs) Against Onartuzumab | Up to approximately 31 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- United States (5):
  - Sarasota, Florida
  - Baltimore, Maryland
  - New York, New York
  - Nashville, Tennessee
  - Houston, Texas
- Pokfulam, Hong Kong
- Singapore, Singapore
- Taiwan (2):
  - Tainan
  - Taipei